CLINICAL TRIAL: NCT06618742
Title: Focal Cryoballoon Ablation for Dysphagia Palliation in Patients with Advanced Esophageal Cancer
Brief Title: Focal Cryoballoon Ablation for Malignant Dysphagia
Acronym: DYS-CBAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Boer (Other)
Responsible Party: Sponsor-Investigator, Laura Boer, Principle Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL84764.000.23
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Dysphagia; Esophageal Cancer; Cryotherapy
Keywords: cryoballoon ablation
MeSH Terms: conditions — Deglutition Disorders; Esophageal Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Cryotherapy — Focal cryoballoon ablation, 1-3 treatments with an interval of 1-3 weeks
  Other Names: cryoballoon ablation

SUMMARY:
Rationale:

Dysphagia is commonly encountered in patients with esophageal carcinoma who are no candidates for treatment with curative intent. It often has a considerable impact on quality of life and can cause malnourishment. Current palliative treatments mainly include esophageal stenting and radiotherapy, but these can be associated with substantial drawbacks such as a high rate of adverse events, fatigue or an untimely/ temporary symptom improvement. Recent studies showed promising results for the use of spray cryotherapy as palliation for dysphagia. Moreover, there are suggestions that cryotherapy has a positive effect on the host's anti-tumor response. However, no data exists on the feasibility, efficacy and safety for cryoballoon therapy in the esophagus. Secondly, cryo-immunologic data in patients with EC is lacking.

Objective:

1. To evaluate the feasibility of cryoballoon ablation in patients with esophageal carcinoma and symptoms of dysphagia. Additionally, efficacy and safety will be assessed.
2. To evaluate the effect of cryoballoon ablation on host's anti-tumor response. Study design: Pilot study, Multi-center Prospective Uncontrolled Intervention

Study Study population: Adult patients (≥18 years) with dysphagia due to incurable esophageal carcinoma Intervention (if applicable): Focal cryoballoon ablation of visible tumor during an upper endoscopy. Cryoballoon ablation will be performed for two cycles of 12 seconds. In total, patients will undergo 3 treatment sessions (range 1-3) with an interval of 1-3 weeks based onthe severity of symptoms reported by the patient.

Main study parameters/endpoints:

* - Feasibility of cryoballoon ablation defined as technical success of the procedure

  * Safety based on incidence of procedure-related serious adverse events
  * Efficacy defined as success rates two weeks after the last cryoablation treatment based on patient reported symptom improvement, and objective evaluation of the esophageal lumen that is free from tumor
* Host's anti-tumor response after cryoballoon ablation based on sequential esophageal tumor biopsies and peripheral blood samples

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years at time of consent
* Histopathologically-confirmed esophageal / gastroesophageal cancer
* Patients in the palliative setting (with or without (future) systemic chemotherapy)
* Dysphagia defined as a score of ≥2 (able to swallow only semi-solids)
* Signed written informed consent

Exclusion Criteria:

* Alternative etiology for dysphagia
* Inability to pass the ultraslim endoscope
* Severe medical comorbidities precluding endoscopy
* Uncorrected coagulopathy
* Prior distal esophagectomy
* Previous esophageal varices
* Expected survival <6 weeks
* Prior radiotherapy for esophageal cancer
* T4b esophageal cancer
* Incapacitated subjects
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome safety | 2 weeks
  Safety based on incidence of all procedure related serious adverse events up to the end of follow-up. The technique is considered to be safe if ≥80% of the procedures is performed without the occurrence of procedure-related serious adverse events.
primary outcome efficacy | 2 weeks
  Efficacy
  * Subjective parameters based on clinical success rate at week 2 after last therapy, using the 5 point Likert dysphagia score (0= no dysphagia, 1= dysphagia to solids, 2= dysphagia to semisolids, 3= dysphagia to liquids, 4= dysphagia to saliva). An improvement of one point is considered as clinical success.
  * Objective parameters:
    * Ability of the diagnostic endoscope to pass
    * Percentage of the diameter of the esophageal lumen that is open/ free from tumor, as assessed by the treating endoscopist and two independent assessors, comparing pre- and post-treatment.
primary outcome feasibility | 1 day
  Feasibility: defined as technical success rates of a full cryotherapy procedure. This includes the ability to pass the scope and the completion of a full circle of freezing and thawing, with the number of cycles needed per site as deemed necessary by the endoscopist. The technique is considered to be feasible if ≥70% of the procedures is technically successful.

SECONDARY OUTCOMES:
secondary outcome efficacy subjective | 2 weeks
  General questions, twice weekly, up to two weeks after last treatment:
  * How do you experience your symptoms now compared to before treatment (0= fully disappeared, 1= symptoms significantly improved, 2= symptoms slightly improved, 3 = symptoms remained the same, 4= symptoms got slightly worse, 5= symptoms got significantly worse)
  * How do you experience your symptoms now compared to yesterday (0= symptoms significantly improved, 1= symptoms slightly improved, 2= symptoms remained the same, 3, symptoms got slightly worse, 4= symptoms got significantly worse)
secondary outcome efficacy subjective | 12 weeks
  Reported outcomes on dysphagia scores twice weekly, up to two weeks after endoscopy, and thereafter at week 6, 8 and 12.
secondary outcome pain | 2 weeks
  Post procedural pain based on twice weekly pain scores up to two weeks after last treatment
  * Pain at the area of the esophageal tumor during meals based on a NRS 0-10 (with 0 indicating no pain and 10 indicating unbearable pain)
  * Pain at the area of the esophageal tumor when not eating/at rest using the same score as above
secondary outcome safety | 12 weeks
  Incidence of all (S)AE's
secondary outcome other palliation | 12 weeks
  Necessity of receiving any other kind of palliation for dysphagia during follow-up
Secondary outcome immunology | 12 weeks
  (Changes in) Host's anti-tumor response after cryoballoon ablation compared to baseline. Analyses on both blood and tissue samples will be performed. Moreover, the peripheral immune response will be compared with the tissue immune response.

CONTACTS AND LOCATIONS:
Locations (1):
- UMCU, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided